CLINICAL TRIAL: NCT05105789
Title: Safe and Healthy Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0790; Protocol Version 5/8/22 (Other: UW Madison); A536756 (Other: UW Madison)
Record Dates: First submitted 2021-10-21; First posted 2021-11-03 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Sars-CoV-2 Infection; COVID-19
Keywords: testing; diagnosis; schools
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- BinaxNOW Test + Lollipop PCR (Experimental): If a symptomatic participant's initial at-school BinaxNOW test was positive, then their study participation is complete after providing the lollipop swab for PCR testing.
  If a symptomatic participant's initial at-school BinaxNOW test was negative, then they will be asked to complete an at-home BinaxNOW test approximately 24 hours later.
  For the at-home BinaxNOW testing, the participant will schedule a follow-up virtual visit with the study coordinator. If they are unable to complete a virtual visit, they will schedule an in-person home visit. They will also be sent home with a BinaxNOW testing kit.
  Interventions: Diagnostic Test: BinaxNOW Test; Diagnostic Test: "Lollipop" swab

INTERVENTIONS:
Diagnostic Test: BinaxNOW Test — diagnostic test for SARS-CoV-2
  Other Names: BinaxNOW COVID-19 Ag Card
Diagnostic Test: "Lollipop" swab — A lollipop swab, is an oral swab to collect saliva, sucked on like a lollipop for 20 seconds.

SUMMARY:
This study will target Madison Metropolitan School District (MMSD) school children ages 4-19 and staff who have not had a previous positive COVID-19 test within the past 3 months. It will enroll children and adults for 1-3 days to explore whether serial "at-home" BinaxNOW testing is feasible and non-inferior to "at school" single PCR testing for the evaluation of symptomatic individuals with a negative initial BinaxNOW. It will also explore whether lollipop swabs are more acceptable and perform as well as nasal swabs with polymerase chain reaction (PCR) testing.

DETAILED DESCRIPTION:
Study Design: This is a quantitative community-based study, conducted in the K-12 setting with school children 4-19 years old, teachers, and staff.

If a participant's initial at-school BinaxNOW test is positive, then they will only complete the lollipop swab for PCR testing. They will NOT do the at-home BinaxNOW test.

If a participant's initial at-school BinaxNOW test is negative, then they will complete both the lollipop swab for PCR testing AND an at-home BinaxNOW test approximately 24 hours later.

If the participant is unwilling or unable to complete the at-home test, they will be presented with a lollipop swab only option.

Aim 1: The investigators will test the hypothesis that serial at-home BinaxNOW testing will be feasible and non-inferior to the single at-school PCR testing program. To do this, the investigators will distribute over-the-counter BinaxNOW antigen tests to volunteer families, and create a protocol to ensure families can perform and report test results accurately to the school.

Two key questions will be addressed:

1. Is 'at-home' BinaxNOW testing feasible for families?
2. Is serial 'at-home' BinaxNOW testing non-inferior to 'at-school' single PCR testing?

Aim 2: The investigators will test the hypothesis that lollipop swabs are more acceptable to individuals and PCR testing is non-inferior to performing PCR on nasal swabs. To test this hypothesis, the investigators will work with MMSD schools to incorporate a lollipop swab for PCR at the time a symptomatic student or staff receives a nasal swab for PCR that is part of the Department of Health Services (DHS) program.

Two key questions will be addressed:

1. Are lollipop swabs more acceptable to individuals when compared to nasal swabs?
2. Will lollipop swabs perform as well as nasal swabs with PCR-based testing?

Hypotheses to be tested:

* Aim 1.1: "At-home" BinaxNOW testing will be feasible for families.
* Aim 1.2: Serial "at-home" BinaxNOW testing is non-inferior to "at school" single PCR testing.
* Aim 2.1: Lollipop swabs are more acceptable to individuals than nasal swabs.
* Aim 2.2: Lollipop swabs will perform as well as nasal swabs with PCR-based testing.

Protocol Amendment 2/4/22 to expand the upper eligible age for children from 14 to 19 years and to recognize the potential supply chain limitations of BinaxNOW tests. If the study team does not have any BinaxNOW tests due to a supply shortage, the BinaxNOW procedures will be dropped and only the lollipop swab will be collected.

Protocol Amendment 5/16/22 extends the study timeline and adds a lollipop swab only option.

ELIGIBILITY:
Inclusion Criteria:

* school children ages 4-19
* MMSD staff
* have at least one symptom of COVID-19
* have not had a positive COVID-19 test in the past 3 months
* will undergo nasal PCR testing at an MMSD elementary school

Exclusion Criteria:

* received a positive COVID-19 test in the past 3 months

Criteria for inclusion in the final study sample:

* Aim 1. Symptomatic participants with a negative at-school BinaxNOW test and nasal PCR results who complete both the lollipop PCR and at-home BinaxNOW tests within 72 hours will be included in the final study sample.
* Aim 2. Symptomatic participants who provide a lollipop swab that is successfully resulted.

Criteria for exclusion in the final study sample:

* Aim 1

  * Missing nasal PCR result
  * Do not successfully complete an at-home BinaxNOW test within 72 hours of the at-school BinaxNOW test
* Aim 2

  * Missing nasal PCR result
  * Missing lollipop PCR result

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Wald, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Community Locations, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Madison Metropolitan School District from October 2021 to May 2023.
Groups:
- COVID-19 Tests: If a symptomatic participant's initial at-school BinaxNOW test was positive, then their study participation is complete after providing the lollipop swab for polymerase chain reaction (PCR) testing.
  If a symptomatic participant's initial at-school BinaxNOW test was negative, then they will be asked to complete an at-home BinaxNOW test approximately 24 hours later.
  For the at-home BinaxNOW testing, the participant will schedule a follow-up virtual visit with the study coordinator. If they are unable to complete a virtual visit, they will schedule an in-person home visit. They will also be sent home with a BinaxNOW testing kit.
  BinaxNOW Test: diagnostic test for SARS-CoV-2
  "Lollipop" swab: A lollipop swab, is an oral swab to collect saliva, sucked on like a lollipop for 20 seconds.
  All participants took the gold-standard Nasal Swab PCR test at school.
Period: Overall Study
Arm/Group | COVID-19 Tests
Started | 100
Number of Participants Who Took the Nasal PCR Test at School | 100
Number of Participants Who Took the Lollipop Test at School | 100
Number of Participants Who Took the BinaxNow Test at School | 100
Number of Participants Who Were Required to Take At-home BinaxNow Test | 79
Number of Participants Who Actually Took the At-home BinaxNow Test | 73
Completed (99 Participants had data from all three COVID-19 tests.) | 99
Not Completed | 1
Not completed — Laboratory's lab collection device damaged | 1

BASELINE CHARACTERISTICS:
Groups:
- COVID-19 Tests: If a symptomatic participant's initial at-school BinaxNOW test was positive, then their study participation is complete after providing the lollipop swab for PCR testing.
  If a symptomatic participant's initial at-school BinaxNOW test was negative, then they will be asked to complete an at-home BinaxNOW test approximately 24 hours later.
  For the at-home BinaxNOW testing, the participant will schedule a follow-up virtual visit with the study coordinator. If they are unable to complete a virtual visit, they will schedule an in-person home visit. They will also be sent home with a BinaxNOW testing kit.
  BinaxNOW Test: diagnostic test for SARS-CoV-2
  "Lollipop" swab: A lollipop swab, is an oral swab to collect saliva, sucked on like a lollipop for 20 seconds.
  All participants took the gold-standard Nasal Swab PCR test at school.
Arm/Group | COVID-19 Tests
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64
  Between 18 and 65 years | 36
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 55
  Male | 43
  Prefer Not to Say | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 79
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 80
  More than one race | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Standard Diagnostic Test Outcomes for BinaxNOW at Home Testing as Compared to Nasal Swab PCR
Description: The primary diagnostic outcome measure will be the negative predictive value (NPV). The kappa values for sensitivity, specificity, positive predictive value (PPV) and NPV of the BinaxNOW at Home testing with respect to PCR nasal swab (gold standard) are reported here.
Time Frame: up to 2 days
Measure: Number (95% Confidence Interval); unit: kappa value in percentage
Units Other Than Participants: At-home Binax tests
Groups:
- BinaxNOW At Home Testing: If a symptomatic participant's initial at-school BinaxNOW test was negative, then they will be asked to complete an at-home BinaxNOW test approximately 24 hours later.
Arm/Group | BinaxNOW At Home Testing
Number analyzed (Participants) | 73
Number analyzed (At-home Binax tests) | 73
kappa value in percentage
  Sensitivity | 100 [44 to 100]
  Specificity | 99 [92 to 100]
  Positive Predictive Value | 75 [30 to 99]
  Negative Predictive Value | 100 [95 to 100]
Statistical Analysis 1: Comparison: BinaxNOW At Home Testing; Negative Predictive Value; Test type: Superiority — One-sample binomial test. Null hypothesis: NPV of BinaxNOW at Home testing is at most 91%. Alternative hypothesis: NPV of BinaxNOW at Home testing is greater than 91%; p = 0.0015, one-sample binomial test; Kappa Co-efficient = 100, 95% CI 2-sided [95 to 100] — binary outcome
Statistical Analysis 2: Comparison: BinaxNOW At Home Testing; Sensitivity H0: Sens-0.99 ≤ 0.05 vs. HA: Sens-0.99 > -0.05; Test type: Non-Inferiority — non-inferiority margin of δ=5% and a sensitivity/specificity of PCR of 99%; p = 0.3308, one-sample binomial test
Statistical Analysis 3: Comparison: BinaxNOW At Home Testing; Specificity H0: Spec-0.99 ≤ 0.05 vs. HA: Spec-0.99 > -0.05; Test type: Non-Inferiority — a non-inferiority margin of δ=5% and a sensitivity/specificity of PCR of 99%; p = 0.0536, one-sample binomial test

2. Primary Outcome: Frequency Table of Gold-Standard Nasal Swab PCR vs Lollipop Swab PCR COVID-19 Test Results
Description: Counts of negative and positive Nasal Swab vs. Lollipop Swab PCR COVID-19 tests with kappa statistical value.
Time Frame: up to 2 days
Population: 1 device did not function properly, 99 participants had data from both test to analyze
Measure: Count of Units; unit: COVID-19 tests
Units Other Than Participants: COVID-19 tests
Groups:
- Negative Nasal Swab PCR: Gold-standard Nasal Swab PCR test, only negative test results reported and compared in this column.
- Positive Nasal Swab PCR: Gold-standard Nasal Swab PCR test, only positive test results reported and compared in this column.
Arm/Group | Negative Nasal Swab PCR | Positive Nasal Swab PCR
Number analyzed (Participants) | 99 | 99
Number analyzed (COVID-19 tests) | 88 | 11
COVID-19 tests
  Lollipop PCR (Negative) | 86 | 0
  Lollipop PCR (Positive) | 2 | 11
Statistical Analysis 1: Comparison: Negative Nasal Swab PCR vs Positive Nasal Swab PCR; Kappa statistics for Nasal Swab PCR vs Lollipop Swab PCR; Test type: Equivalence — Concordance between the PCR test results will be evaluated by calculating the Kappa statistic which will be reported along with corresponding two-sided 95% confidence interval. The nonparametric bootstrap technique will be used to construct the confidence interval. A kappa statistic of >0.95 will be considered as sufficient to define lollipop swab test non-inferior to the gold-standard PCR testing of nasal swabs; Kappa Co-efficient = 0.91, 95% CI 2-sided [0.78 to 1.00]

3. Primary Outcome: Standard Diagnostic Test Outcomes for Lollipop Swab PCR Testing as Compared to Nasal Swab PCR
Description: The kappa values for sensitivity, specificity, positive predictive value (PPV) and NPV of the Lollipop Swab PCR with respect to PCR nasal swab (gold standard) are reported here.
Time Frame: up to 2 days
Population: 1 device did not function properly, 99 participants had data from both test to analyze
Measure: Number (95% Confidence Interval); unit: kappa value in percentage
Units Other Than Participants: COVID-19 tests
Groups:
- Lollipop Swab PCR Testing: A lollipop swab, is an oral swab to collect saliva, sucked on like a lollipop for 20 seconds. Participants used the lollipop swab at school.
Arm/Group | Lollipop Swab PCR Testing
Number analyzed (Participants) | 99
Number analyzed (COVID-19 tests) | 99
kappa value in percentage
  Sensitivity | 100 [74 to 100]
  Specificity | 98 [92 to 99]
  Positive Predictive Value | 85 [58 to 96]
  Negative Predictive Value | 100 [96 to 100]
Statistical Analysis 1: Comparison: Lollipop Swab PCR Testing; Sensitivity H0: Sens-0.99 ≤ 0.05 vs. HA: Sens-0.99 > -0.05; Test type: Non-Inferiority — a non-inferiority margin of δ=5% and a sensitivity/specificity of PCR testing of 99%; p = 0.2010, one-sample binomial test
Statistical Analysis 2: Comparison: Lollipop Swab PCR Testing; Specificity H0: Spec-0.99 ≤ 0.05 vs. HA: Spec-0.99 > -0.05; Test type: Non-Inferiority — non-inferiority margin of δ=5% and a sensitivity/specificity of PCR testing of 99%; p = 0.0705, one-sample binomial test

4. Primary Outcome: Number of Successfully Completed At-home Tests
Description: Feasibility of 'at-home' BinaxNOW testing will be determined by number of successfully completed at-home tests. At-home test taking will be monitored by study team remotely (via zoom or similar).
Time Frame: up to 24 hours
Measure: Count of Units; unit: at home COVID-19 tests
Units Other Than Participants: at home COVID-19 tests
Groups:
- At Home BinaxNOW Test: For the at-home BinaxNOW testing, the participant will schedule a follow-up virtual visit with the study coordinator. If they are unable to complete a virtual visit, they will schedule an in-person home visit. They will also be sent home with a BinaxNOW testing kit.
  BinaxNOW Test: diagnostic test for SARS-CoV-2
Arm/Group | At Home BinaxNOW Test
Number analyzed (Participants) | 79
Number analyzed (at home COVID-19 tests) | 73
at home COVID-19 tests | 73

5. Primary Outcome: Percent of Participants Who Answer 'Yes' When Asked if Lollipop Swabs Are More Acceptable Than Nasal Swabs
Description: To address the acceptability of lollipop swabs vs nasal swabs, the study team will ask participants a binary question: Are lollipop swabs more acceptable to participants when compared to nasal swabs? Yes/No.
Time Frame: up to 1 day
Measure: Count of Participants; unit: Participants
Groups:
- COVID-19 Tests: "Lollipop" swab: A lollipop swab, is an oral swab to collect saliva, sucked on like a lollipop for 20 seconds.
  vs. the gold-standard nasal swab PCR experience.
Arm/Group | COVID-19 Tests
Number analyzed (Participants) | 100
Participants | 92

ADVERSE EVENTS:
Time Frame: Adverse events were collected after consent was signed and until they completed study procedures during the school visit or during the Binax Now visit (up to 5 days)
Groups:
- COVID-19 Tests: If a symptomatic participant's initial at-school BinaxNOW test was positive, then their study participation is complete after providing the lollipop swab for PCR testing.
  If a symptomatic participant's initial at-school BinaxNOW test was negative, then they will be asked to complete an at-home BinaxNOW test approximately 24 hours later.
  For the at-home BinaxNOW testing, the participant will schedule a follow-up virtual visit with the study coordinator. If they are unable to complete a virtual visit, they will schedule an in-person home visit. They will also be sent home with a BinaxNOW testing kit.
  BinaxNOW Test: diagnostic test for SARS-CoV-2
  "Lollipop" swab: A lollipop swab, is an oral swab to collect saliva, sucked on like a lollipop for 20 seconds.
Arm/Group | COVID-19 Tests
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

LIMITATIONS AND CAVEATS:
Some limitations and caveats of this study include:

* Difficulty enrolling participants because parents were not allowed into the school building for the informed consent procedure.
* The outdoor consenting procedure became more difficult, and at times impossible, during extreme cold, or rainy weather days.
* School holidays during COVID surges, and the COVID Clinic's proximity and lack of cooperation also created limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT05105789/Prot_SAP_000.pdf